CLINICAL TRIAL: NCT03685071
Title: Prognostic Value of Complete Blood Count in Children Suffering of Severe Infections in Pediatric Care Unit
Brief Title: Prognostic Value of Complete Blood Count in Severe Infections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Heshmat, principal investigator, Assiut University
Other Study IDs: PVCCSFSI
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Infection Systemic
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: role of CBC as prognostic tool in sepsis. — Our study will be conducted on children who admitted to PICU in Assuit University Hospital .CBC parameters as TLC , platelet count , and Hb will be evaluated at time of admission , another CBC will be done at 5th day and another one at day of discharge or last one before death.
  * patients will be classified into three groups according to the outcome(discharge, mortality and has morbidity sequel.)
  * correlation between the outcome and CBC will be done.

SUMMARY:
Sepsis is a leading cause of hospitalization in pediatric intensive care units, In the last decade, a series of initiatives were implemented that aim not only to improve the understanding of sepsis and the clarity of concepts related to this condition but also to reduce morbidity and mortality due to sepsis through earlier diagnosis and initiation of antibiotic therapy as well as through the provision of specific guidelines for the treatment of pediatric sepsis. Despite these measures and the lower mortality from sepsis in children compared to adult patients, the impact of sepsis in the pediatric population remains high.

DETAILED DESCRIPTION:
According to the World Health Organization, sepsis remains a leading cause of death in infants and children in developed and developing countries.Some prognostic scoring systems with performance status, clinical symptoms, and biochemical parameters help to guide accurate prediction of the prognosis, such as the acute physiology and chronic health evaluation (APACHE), yet are considered too complex for general clinical use. Therefore, the prediction of clinical events with laboratory parameters, including complete blood cell count (CBC), has become an increased focus of research.

Accumulating evidence indicates that the CBC is an effective predictor of prognosis and mortality in many disease states, including hematological disease, neoplasms, and diseases of the circulatory system severe infections. Therefore, nonspecific changes in the CBC in critically ill patients could be considered a key prognostic factor in the evaluation of survival prediction in these patients .

According , it is possible that the CBC could be used as a predictor of survival in severe infections patients. The complete blood count (CBC) , a five-cell automated differential count and a reflex manual differential count (when required by protocol) and is one of the most frequently ordered admission laboratory tests.

In practice, it is a routine ingredient of all hospital admission orders - a complete blood count is done for our medical , surgical admissions and the same is true at most institutions . it is known that the white blood cell count do predict disease severity and mortality risk. For example, elevated WBC counts predict a worse prognosis in patients with severe infections in pediatric intensive care unit ,Further, this test provides direct management guidance in common circumstances, e.g., infection.

The CBC describes the number and morphology of over 40 different cells. Disagreement exists regarding the clinical significance of many of these observations. And only a few components of the manual differential, e.g., nucleated red blood cells and lymphocytes, have been quantitatively evaluated to determine their prognostic significance. But these two observations have not been examined to determine their independent contributions to mortality predictions when taken in conjunction with their accompanying CBC observations. .

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 18 years and > one month .
2. patient presented with sepsis defined as suspected source of infection (we defined sepsis using predetermined international sepsis definitions as clinical syndrome with both infection and a systemic inflammatory response) .
3. Abnormal leukocyte count >12×109 /cmm or<4 × 109/cmm or>10% immature form.
4. patients presented with secondary organ dysfunction.

Exclusion Criteria:

1. Age more than 18 years and age less than one month.
2. patient with active bleeding.
3. patient who had used anti platelet drugs .
4. patient not diagnosed sepsis or septic shock.

Ages: 30 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: * patients will be classified into three groups according to the outcome(discharge, mortality and has morbidity sequel.)
  * Correlation between the outcome and blood culture will be done.
  * correlation between the out come AndCRPwill be done.
  * Then another correlation between the outcome and CBC will be done.
  * Comparison between the two previous correlations will be done to detect if CBC alone can predict the outcome of the patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
prognosis of outcome in patients suffering from severe infections in PICU by using CBC . | one year
  Complete blood count in children aged between one month and 18 years suffering of infections is enough as prognostic tool and predict the out come or not enough and more investigation will be required by correlation between CBC and the outcome of patients dead or discharge or morbid sequel.

CONTACTS AND LOCATIONS:
Overall Officials: doaa heshmat, Principal Investigator — Assiut University